CLINICAL TRIAL: NCT06496737
Title: Effects of Moderate-Intensity Interval Training (MIIT) on Mental Toughness, Sports Motivation, Athlete Burnout, Perceived Stress, Unforced Errors and Performance of Competitive Badminton Players in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wu Jiarun (Other)
Responsible Party: Sponsor-Investigator, Wu Jiarun, student, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Li Chongwei
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Burnout，Motivation，Stress，Mental Toughness
Keywords: Burnout，motivation，stress and mental toughness of badminton players
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: The 171 people tested were randomly divided into 3 groups of 57 each during the intervention phase, with two groups carrying out a intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Interval Training (MIIT) (Experimental): Moderate-Intensity Interval Training (MIIT) is developed by university badminton coaches
  Interventions: Behavioral: Moderate-Intensity Interval Training (MIIT)
- High-Intensity Interval Training (HIIT) (Experimental): High-Intensity Interval Training (HIIT) is developed by university badminton coaches
  Interventions: Behavioral: High-Intensity Interval Training (HIIT)

INTERVENTIONS:
Behavioral: Moderate-Intensity Interval Training (MIIT) — Moderate-Intensity Interval Training (MIIT) is developed by university badminton coaches, three times a week for 12 weeks
  Arms: Moderate-Intensity Interval Training (MIIT)
Behavioral: High-Intensity Interval Training (HIIT) — High-Intensity Interval Training (HIIT) is developed by university badminton coaches, three times a week for 12 weeks
  Arms: High-Intensity Interval Training (HIIT)

SUMMARY:
The objective of this observational study was to assess whether moderate intensity training (MIIT) intervention has positive effects on Mental Toughness, Sports Motivation, Athlete Burnout and Perceived Stress of badminton players in Yunnan Province. And reduce the error rate of badminton players

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants were between the ages of 18 to 30

  2. Male or female

  3. At least 3 years' experience in amateur badminton training. This includes current players who are training with the Province badminton team. Or has been selected by the Kunming badminton team in Yunnan Province. Or have participated in domestic or foreign provincial, municipal or higher's competitions.

Exclusion Criteria:

- 1. Participants who are currently injured. 2. Participants who have not participated in any provincial badminton competition.

3. Participants who refuse to give consent to participate in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 171 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Reduce the error rate of badminton players | week 12
  The error rate will be recorded by a professional video camera team, recorded and counted by the teaching assistant team, and calculated and analyzed by the head coach

SECONDARY OUTCOMES:
Change from mental toughness questionnaire (MTQ) | week 12
  Sports Mental Toughness Questionnaire (SMTQ; Clifford et al., 2007) consisted of 14 questions to assess the three dimensions of confidence, persistence and control, and was scored using the 4-point Likert scale. The results of confirmatory factor analysis (CFA) show that the model fits well, and the specific indicators are as follows: Chi-square value χ² = 120.50, df = 71, p < 0.001, comparative fitting index (CFI) was 0.93, value-added fitting index (TLI) was 0.91, root mean square approximation (RMSEA) was 0.05, and standardized mean square residual (SRMR) was 0.06. These results indicate that SMTQ has good structural validity and reliability, and is suitable for evaluating the mental toughness of athletes.
Change from athlete burnout questionnaire (ABQ) | week 12
  Athlete Burnout Questionnaire (ABQ; Marie et al., 2010) consisted of 15 questions assessing three dimensions of emotional and physical exhaustion, reduced exercise value, and exercise isolation using a 5-point Likert scale. The results of confirmatory factor analysis (CFA) show that the model fits well, and the specific indicators are as follows: Chi-square value χ² = 178.30, df = 87, p < 0.001, comparative fitting index (CFI) was 0.92, value-added fitting index (TLI) was 0.90, root mean square approximation (RMSEA) was 0.06, and standardized mean square residual (SRMR) was 0.05. These results indicate that ABQ has good structural validity and reliability and is suitable for evaluating the degree of burnout in athletes.
Change from sport motivation scale-6 (SMS-6） | week 12
  Sport Motivation Scale-6 (SMS-6; Mallet et al., 2007) consisted of 24 questions assessing three main dimensions: intrinsic motivation, extrinsic motivation, and unmotivation, scored using a 7-point Likert scale. The total Cronbach's Alpha value of the questionnaire was 0.85. The results of confirmatory factor analysis (CFA) showed that the model was well fitted, with specific indicators as follows: Chi-square value χ² = 320.75, df = 216, p < 0.001, comparative fitting index (CFI) was 0.93, value-added fitting index (TLI) was 0.92, and root-mean-square error approximation (RMSEA) was 0.05. These results indicate that SMS-6 has good structural validity and reliability and is suitable for evaluating athletes' motivation.
Change from Perceived Stress Questionnaire（PSQ） | week 12
  Perceived Stress Questionnaire (PSQ; Sanz et al., 2001) consisted of 30 questions to assess subjective feelings of stress, scored using a 4-point Likert scale. The results of confirmatory factor analysis (CFA) show that the model fits well, and the specific indicators are as follows: Chi-square value χ² = 450.65, df = 400, p < 0.001, comparative fitting index (CFI) was 0.91, value-added fitting index (TLI) was 0.90, root mean square approximation (RMSEA) was 0.04, and standardized mean square residual (SRMR) was 0.05. These results indicate that PSQ has good structural validity and reliability, and is suitable for assessing the subjective stress perception of individuals.
Heart rate variability (HRV) Heart rate variability (HRV) | week 12
  HRV data were collected using a heart rate variability (HRV) analyser.
Blood oxygen saturation (SaO2) | week 12
  Blood oxygen saturation (SaO2) data were collected using an oxygen saturation tester.

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Sains Malaysia, Kota Bharu, Kelantan, Malaysia